CLINICAL TRIAL: NCT04671589
Title: Antidote for Valproic Acid Toxicity: a New Indication for Meropenem Antibiotic. A Randomized Placebo-controlled Trial
Brief Title: Antidote for Valproic Acid Toxicity: a New Indication for Meropenem Antibiotic.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mabaret Al-Asafara Hospitals (Network)
Responsible Party: Principal Investigator, Nancy Mohamed, Clinical pharmacist, Mabaret Al-Asafara Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N2014
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Drug Toxicity
Keywords: Valproic acid toxicity - Meropenem - Antidote
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Meropenem; Palliative Care; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meropenem (Experimental): Meropenem 1 gram intravenous every 8 hours
  Interventions: Drug: Meropenem Injection
- Placebo (Placebo Comparator): Placebo intravenous every 8 hours
  Interventions: Drug: Meropenem Injection

INTERVENTIONS:
Drug: Meropenem Injection — Administration Intravenous meropenem 1gram every 8 hours together with standard care;
  .
  Other Names: Supportive care as fluids and securing airway if needed

SUMMARY:
Acute Valproic acid (VPA) toxicity is an emergency condition which may commonly present with central nervous system (CNS) depression(5). In mild poisoning, associated with VPA ingestions of 200 mg/kg, sedation and lethargy commonly occur(6); while in severe VPA poisoning associated with ingestions of 400 mg/kg or more, life threatening events are likely to occur as respiratory depression, metabolic acidosis, encephalopathy, hemodynamic instability, and cerebral edema which may progress to coma and even death -if not treated promptly. Supportive care along with early gastric decontamination using activated charcoal (AC) (which may only be given if patient presented early after ingestion), in addition to intravenous (IV) administration of Levocarnitine (L-Carnitine) and ensuring adequate airway protection are the cornerstone of treatment, but there remains no drug listed as a specific antidote for acute VPA intoxication. Carbapenem antibiotics augment the clearance of VPA through suppressing its enterohepatic recirculation, as they inhibit the acylpeptide hydrolase enzyme responsible for the reabsorption of the hydrolyzed valproate back to VPA active molecule. Taking advantage of this well-established drug-drug interaction between VPA and carbapenems resulting in significant drop of VPA serum concentration during concomitant use, we propose that administration of meropenem (member of carbapenems group) will prove effectiveness in managing VPA toxicity by achieving lower plasma levels of VPA and/or enhanced alertness; compared with standard care.

DETAILED DESCRIPTION:
JUSTIFICATION AND SIGNIFICANCE:

Valproic acid (VPA) -a branched chain carboxylic acid- introduced by the Food and Drug Administration in 1978 for the treatment of seizure disorders(1). In the following years, VPA gained further approved indications to treat bipolar and behavioral disorders(2), migraine prophylaxis(3) as well as other psychiatric indications(4).The growing use of VPA and its availability resulted in increased prevalence of VPA overdoses(5,6). The rising incidence of acute VPA toxicity is either resulting from suicidal attempts, accidental ingestions, or following VPA dose increments to achieve the desired therapeutic effect(7). Acute VPA toxicity is an emergency condition which may commonly present with central nervous system (CNS) depression(5). In mild poisoning, associated with VPA ingestions of 200 mg/kg, sedation and lethargy commonly occur(6); while in severe VPA poisoning associated with ingestions of 400 mg/kg or more, life threatening events are likely to occur as respiratory depression, metabolic acidosis, encephalopathy, hemodynamic instability, and cerebral edema which may progress to coma and even death -if not treated promptly(5,8). Serum VPA concentration is the most functional tool in diagnosing and determining the severity of toxicity. Supportive care along with early gastric decontamination using activated charcoal (AC) (which may only be given if patient presented early after ingestion), in addition to intravenous (IV) administration of Levocarnitine (L-Carnitine) and ensuring adequate airway protection are the cornerstone of treatment, but there remains no drug listed as a specific antidote for acute VPA intoxication(5,9).

Carbapenems are a group of β-lactam antibiotics with a growing need to use in the empiric and definitive treatment, due to the emerging resistance to antibiotics(10). A multitude of case reports(11-13), retrospective observational studies(14-19) and reviews(20-22) demonstrated that combined use of VPA and carbapenem antibiotics -mainly meropenem (16)(23)- is associated with a potential drug interaction that can significantly decrease VPA serum concentration(24). One retrospective trial included 36 patients concluded that VPA mean ± SEM serum concentration dropped from 50.8 ± 4.5 µg/mL to 9.9 ± 2.1 µg/mL(P < .001) following meropenem administration with a mean decrease of 82.1% ± 2.7%(18), while a recent prospective observational trial determined that the mean drop in serum VPA level was 80% ranging from(49%-99%)(23). However, despite VPA toxicity with fatal events being reported for over 20 years, only a few case reports documented successful intentional use of meropenem as an antidote for VPA poisoning(25-27). To date, no randomized-controlled trials were conducted.

Specific aims: Determine if meropenem is effective in treating acute VPA toxicity, manifested by achieving reduced VPA plasma levels and/or enhanced mentation.

Hypothesis: Administration of meropenem combined with standard care is effective in managing VPA intoxication, affirmed by providing lower serum VPA concentrations and/or better level of consciousness; in contrast to standard care alone.

Background: VPA is an antiepileptic drug that has psychiatric indications as well(28). VPA acute intoxication is a critical condition listed among fatal pharmaceutical exposures, with CNS toxicity being the most common manifestation and may progress to respiratory depression and/or coma(5). In 2018, the American Association of Poison Control Centers (AAPCC) Toxic Exposure Surveillance System (TESS) database reported 7699 VPA exposures, of which: 2079 were treated in health care facilities, 87 resulted in major toxicity, and 19 resulted in deaths(29). These data denote that VPA poisoning is becoming an area of growing concern among toxicologists.

Supportive care and ensuring adequate airway protection are the cornerstone of treatment; yet, no drug specified as an antidote for managing VPA intoxication(5). Carbapenem antibiotics augment the clearance of VPA through suppressing its enterohepatic recirculation, as they inhibit the acylpeptide hydrolase enzyme responsible for the reabsorption of the hydrolyzed valproate back to VPA active molecule(21). Taking advantage of this well-established drug-drug interaction between VPA and carbapenems resulting in significant drop of VPA serum concentration during concomitant use(15,17,23), we propose that administration of meropenem (member of carbapenems group) will prove effectiveness in managing VPA toxicity by achieving lower plasma levels of VPA and/or enhanced alertness; compared with standard care.

Research design and methodology:

Operational definitions of research variables:

VPA toxicity: Ingestion of VPA, at doses higher than 60 mg/kg/day, with a serum VPA concentration above the therapeutic threshold of 100 µg/mL and/or altered sensorium.

Standard care: Encompasses supportive care: administration of IV fluids, endotracheal intubation for securing airway in patients with altered sensorium, benzodiazepines should be administered only if seizures occur and L-carnitine 100 mg/kg IV in cases of hyperammonemia.

Primary outcome: Evaluate serum VPA concentrations among the two study groups. Secondary outcome: Assess patients level of consciousness according to the Glasgow Coma Scale (GCS) among the placebo and treatment groups.

Study Design and Location: This is a multicentered, randomized (1:1), double blinded, placebo controlled study where eligible patients will be randomly assigned into two groups using simple random sample technique, each patient will either receive: IV meropenem 1gram every 8 hours together with standard care; or placebo along with standard care. Computer generated random number tables, will be used to allocate patients to either treatment or placebo groups. We will make the participant and the assessing physician unaware of the treatment. The study will be conducted in three poison control centers (PCC) in Egypt: (1) poison control center of Ain Shams university hospitals; (2) poison control center of Alexandria university hospitals; (3) poison control center of Tanta university hospitals. We will obtain their institutional review board and/or ethics committee approval to conduct the study protocol prior to study initiation.

Interventions and Monitoring: Serial VPA serum concentrations to be assessed every two to four hours until a steady significant declined level is noted, while neurological status assessment of patients will be performed according to the GCS three times daily.

Sample Size & Power: Based on VPA toxicity levels, mean VPA serum level of 378.3 mg/mL ± 310.2 mg/mL were reported(7), following meropenem administration, the mean drop in serum VPA level was 80%(18,23). Owing to this data, we estimated that a minimum of 48 patients will be needed to confirm this effect (α= 5% and power of 90 %).

Study duration: Reviewing annual reports of PCCs in Egypt, a single PCC received 44 cases of VPA toxicity throughout the year 2011(30). Hence, an estimated one-year duration will be sufficient to conduct our study over three PCCs in Egypt.

Proposed statistical analysis: Data will be presented as mean ± standard deviation or median with interquartile range. Differences between the two groups will be tested using independent sample t-test or Mann-Whitney U-test. Univariate analysis for comparing different demographic data between meropenem group and placebo group using Chi square test and t-test as applicable, Linear regression will be used to adjust for confounders. The analysis will be carried out according to the intention to treat principle.

Differences will only be considered significant at P <0.05 and statistical analysis will be performed using the Stata statistical software, version 16.0.

Study Limitations: 1) VPA overdoses may occur among patients with history of epilepsy. Meropenem is a drug that possess seizure potential, but mainly seizures were reported in patients with history of epilepsy and patients with declined renal function. Meanwhile, overall seizure rate being 0.7% among immunocompetent patients (24). Meropenem dosage reduction is recommended in patients with advanced age and/or patients with renal impairment.

Compliance to the recommended dosage regimens in addition to bedside digital electroencephalogram (EEG) tracings will be urged in epileptic patients.

2) The results of this study would only apply to patients with the study inclusion criteria, further studies should be conducted to cover the excluded criteria population.

Anticipated results: Meropenem with standard care will exhibit effectiveness in VPA toxicity treatment, by achieving lower mean serum concentrations of VPA and/or higher median GCS denoting improved sensorium; when compared with standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with VPA toxicity will be included if aged 18 years or more. The patient himself/herself should provide informed consent; a family member may take place only if there is an altered mentation that may hinder such procedure.

Exclusion Criteria:

* Patients will be excluded if presenting one hour following VPA ingestion and were administered AC for gastric decontamination, as it may decrease VPA bioavailability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate serum Valproic acid concentrations among the two study groups. | 1 year
  Plasma level of valproic acid

SECONDARY OUTCOMES:
Assess patients level of consciousness according to the Glasgow Coma Scale (GCS) among the placebo and treatment groups. Assess patients level of consciousness according to the Glasgow Coma Scale (GCS) among the placebo and treatment groups. | 1 year
  Glasgow coma scale ranging from 3 (not responsive) to 15 (responsive)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Ahmed, MSc, Principal Investigator — Clinical pharmacist
Locations (1):
- Alexandria University hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No